CLINICAL TRIAL: NCT02765880
Title: Time,Self and Spontaneous Mental Activities in Patients With Psychotic Disorders
Acronym: Self and Time
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: not enough patients avalaible
Sponsor: University Hospital, Strasbourg, France (Other)
Collaborators: Fondation pour la Recherche Médicale (FRM) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 6366
Record Dates: First submitted 2016-04-15; First posted 2016-05-09 (Estimated); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Schizophrenia; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy volunteer (Experimental)
  Interventions: Other: fMRI; Other: EEG
- Patients with schizophrenia (Experimental)
  Interventions: Other: fMRI; Other: EEG
- Patient with bipolar disorder (Experimental)
  Interventions: Other: fMRI; Other: EEG

INTERVENTIONS:
Other: fMRI — Connectivity between the areas related to information processing over time and the areas activated during the rest activity. We will verify whether the activation anomalies observed during time tasks predict anomalies in spontaneous activity dynamics.
Other: EEG — link between EEG response anomalies related to information processing over time and response anomalies recorded during rest activity. We will check whether anomalies in EEG oscillatory responses during time tasks predict anomalies during the rest task.

SUMMARY:
The main purpose of the study is to examine to which extent abnormalities in the dynamics of neural activities observed in patients with psychosis is related to difficulties at ordering simple visual stimuli and/or personal events.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* Affiliation to a social security insurance
* Written consent given
* Only for patient : DSM criteria for schizophrenia or bipolar disorder

Exclusion Criteria:

* Addiction problem
* Invalidating visual sensory problems
* Neurological history
* Pregnancy or breastfeeding
* Legal safeguard
* Participation in another clinical trial
* Contraindication to MRI

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2017-03-16 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Abnormalities in connectivity during order judgement tasks will be taken as seeds to check whether they account for abnormalities in connectivity at rest, by means of mathematic modelization | After study completion (2 years)

SECONDARY OUTCOMES:
Evaluation of the brain' functional coupling dynamics over time (how neuronal networks and connectivity change over time) during rest. | After study completion (2 years)
- Evaluation of the brain' functional coupling dynamics over time (how neuronal networks and connectivity change over time) during time ordering. | After study completion (2 years)
Comparison of patients with schizophrenia vs. bipolar disorder | During fMRI and EEG sessions

CONTACTS AND LOCATIONS:
Overall Officials: Anne GIERSCH, Principal Investigator — Strasbourg's University Hospitals - INSERM 1114 Unit
Locations (1):
- Service de psychiatrie, Strasbourg, France